CLINICAL TRIAL: NCT07132606
Title: Serum Histone Succinylation: A Predictive Biomarker for Malignant Solid Tumors
Brief Title: The Predictive Value of Serum Histone Succinylation in Malignant Solid Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: Yinghua Ji (Other)
Responsible Party: Sponsor-Investigator, Yinghua Ji, Doctor, The First Affiliated Hospital of Xinxiang Medical College
Organization: The First Affiliated Hospital of Xinxiang Medical College (Other)
Other Study IDs: CHASE 016; Chase 016 (Other: The First Affiliated Hospital of Xinxiang Medical College)
Record Dates: First submitted 2025-07-15; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Malignant Tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 500 patients with malignant solid tumors: Aged ≥18 years, regardless of sex； Histologically or cytologically confirmed malignant solid tumors requiring subsequent anticancer therapy

SUMMARY:
In recent years, advances in protein post-translational modification (PTM) research have revealed histone succinylation as a novel epigenetic modification mechanism critically involved in tumor initiation, progression, and prognosis. Succinylation alters protein physicochemical properties and functions, thereby modulating cellular metabolism, proliferation, and apoptosis. Aberrant histone succinylation in tumor cells demonstrates significant correlations with tumor type, staging, and clinical outcomes, offering new avenues for early cancer diagnosis.

This project utilizes blood serum samples to quantify histone succinylation levels through modification-specific antibody-based detection. Integrated with clinical data, this approach enables early, rapid, and accurate pan-cancer diagnosis, achieving tumor screening via a single-tube blood test. It represents a paradigm shift in precision oncology from "gene-driven" to "epigenetic-metabolic-driven" early detection.

DETAILED DESCRIPTION:
Primary Objective To evaluate differential expression of serum histone succinylation between malignant solid tumor patients and healthy controls, thereby validating its early detection value.

Secondary Objectives

To determine correlations between serum histone succinylation levels and:

Tumor types Tumor stages

To statistically analyze associations of serum histone succinylation with:

Therapeutic efficacy (surgical intervention, radiotherapy, systemic therapy) Clinicopathological variables

ELIGIBILITY:
Inclusion Criteria:

Case Group:

* Aged ≥18 years, regardless of sex；
* Histologically or cytologically confirmed malignant solid tumors requiring subsequent anticancer therapy；

Control Group:

* Aged ≥18 years, regardless of sex；
* Non-cancer participants enrolled through health screenings；

Exclusion Criteria:

* Pregnant individuals；
* Individuals with serious mental disorders or communication barriers；
* Other conditions deemed by investigators to contraindicate study participation；

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with malignant tumors and healthy individuals
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the positive rate of serum histone succinylation in patients with malignant solid tumors | 2025.08.01-2026.12.31
  Evaluate the positive rate of serum histone succinylation in malignant solid tumor patients versus healthy individuals through Western blot analysis, quantify the percentage difference between the two groups, and thereby validate its potential for early cancer screening

SECONDARY OUTCOMES:
Define the relationship between histone succinylation modifications in serum and different tumor types as well as tumor staging | 2025.08.01-2026.12.31
  Analyze the relationship between histone succinylation modifications in serum and therapeutic efficacy (specifically surgery, radiotherapy, and systemic therapy)。

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF
Time Frame: 2025.08.01-2026.12.31

DOCUMENTS (1):
  • Study Protocol (2025-07-19): https://cdn.clinicaltrials.gov/large-docs/06/NCT07132606/Prot_000.pdf